CLINICAL TRIAL: NCT00126776
Title: VISN 23 Lung Disease Self Management/Case Management Program
Brief Title: Veterans Integrated Service Network (VISN) 23 Lung Disease Self Management/Case Management Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Kathryn Rice MD, Minneapolis VA Medical Center
Organization: VA Midwest Health Care Network (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VISN 23 PC-SI 0401
Record Dates: First submitted 2005-08-03; First posted 2005-08-04 (Estimated); Results first posted 2009-08-25 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary disease; case management; self management
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Case Management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): CAse/self management for COPD
  Interventions: Behavioral: case management
- 2 (Other): usual care
  Interventions: Behavioral: usual care

INTERVENTIONS:
Behavioral: case management — case/self management for COPD vs usual care
  Arms: 1
Behavioral: usual care — usual care for COPD
  Arms: 2

SUMMARY:
The purpose of this study is to determine if a program of self management and case management reduces hospitalizations and urgent care visits for patients with chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
Study design and plan:

This is a one-year, 5-site randomized trial. High-risk patients will be randomized to usual care or a case/self management intervention. The frequency of urgent care visits or admission to a hospital for COPD will be compared.

Study procedures: visit 1 Patient informed consent will be obtained prior to patient participation in the trial.

Patients will also sign a release of information form to obtain outside records of COPD admissions or urgent care visits.

Demographic data, inclusion/exclusion data, medications and problem list will be obtained.

Post-albuterol forced expiratory volume in 1 second (FEV1) and forced vital capacity (FVC) will be performed using calibrated spirometers in accordance with guidelines established by the American Thoracic Society. A uniform set of nomograms (NHANES III) will be used at all sites. The best of three efforts will be defined as the highest FEV1 and the highest FVC obtained on any of the three blows (even if not from the same curve with a maximum of 5 attempts).

Patients who meet all above criteria and who agree to participation will be randomized to usual care or the case/self management intervention, by means of sealed sequentially numbered envelopes at each site.

Patients who are randomized to case/self management intervention will receive 1-2 hours of education (appendix 1). These patients will be given instructions for self-management of exacerbation and a telephone care contact number. Coordinators will confirm that the patient has been instructed about, and is in possession of, standard pharmacologic treatment of exacerbation, including a 10 day supply of oral prednisone and an oral antibiotic. Prednisone dose regimens and specific antibiotics will be determined by the site PI according to local sensitivities and practice patterns, with access to current disease management recommendations and information.

Study procedures: treatment period All patients will be contacted by telephone every 6 weeks by a blinded centralized study staff member who will inquire about interim urgent care visits and hospitalizations and COPD exacerbations according to a scripted case report form.

Patients in the intervention arm will be contacted by the site coordinator monthly to reinforce educational principles and assist patients with disease management questions or concerns.

Study procedures: end of trial At the end of one year quality of life scores (SF36 and St. George's Respiratory Questionnaire, a VISN 23 patient satisfaction survey, and a brief questionnaire regarding current influenza and pneumococcal vaccination status, smoking status, and average number of minutes of exercise per day will be mailed to all patients.

ELIGIBILITY:
Inclusion Criteria:

One or more of the following:

* Hospital admission for COPD within the prior year
* Unscheduled visit for COPD within the prior year
* Home oxygen use for COPD
* Systemic steroid use for COPD within the prior year
* Post bronchodilator FEV1 < 70% predicted
* Post bronchodilator FEV1/FVC < 70% predicted

Exclusion Criteria:

* Any unstable medical condition that would preclude effective participation in the study, or which would be expected to reduce life expectancy to < 1 year
* Inability to contact patient by telephone

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 743 (Actual)
Dates: Start 2004-07; Primary Completion 2007-12 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn L Rice, MD, Principal Investigator — Minneapolis Veterans Affairs Medical Center; Naresh Dewan, MD, Principal Investigator — VA Nebraska Western Iowa Health Care System
Locations (5):
- United States (5):
  - Des Moines VA, Des Moines, Iowa
  - IA City VA, Iowa City, Iowa
  - Minneapolis VAMC, Minneapolis, Minnesota
  - Omaha VAMC, Omaha, Nebraska
  - Sioux Falls VAMC, Sioux Falls, South Dakota

REFERENCES:
- [Derived] Rice KL, Dewan N, Bloomfield HE, Grill J, Schult TM, Nelson DB, Kumari S, Thomas M, Geist LJ, Beaner C, Caldwell M, Niewoehner DE. Disease management program for chronic obstructive pulmonary disease: a randomized controlled trial. Am J Respir Crit Care Med. 2010 Oct 1;182(7):890-6. doi: 10.1164/rccm.200910-1579OC. Epub 2010 Jan 14. PMID 20075385

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruited by VA mailing lists July 2004-June 2006
Groups:
- Disease Management for COPD: disease management for COPD
- Usual Care: usual care
Period: Overall Study
Arm/Group | Disease Management for COPD | Usual Care
Started | 372 | 371
Completed | 372 | 371
Not Completed | 0 | 0
Not completed — follow up complete on all patients | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Disease Management for COPD | Usual Care | Total
Number analyzed (Participants) | 372 | 371 | 743
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 127 | 103 | 230
  >=65 years | 245 | 268 | 513
Age Continuous [Mean (Standard Deviation); unit: years] | 69.1 (9.4) | 70.1 (9.7) | 70.1 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 363 | 365 | 728
Region of Enrollment [Number; unit: participants]
  United States | 372 | 371 | 743

OUTCOME MEASURES:

1. Primary Outcome: Hospitalization or Emergency Department Visit for COPD
Time Frame: 1 yr
Reporting Status: Not Posted

2. Secondary Outcome: All Cause Hospitalizations
Time Frame: 1 year
Reporting Status: Not Posted
Measure: Mean (95% Confidence Interval)

3. Secondary Outcome: Quality of Life
Time Frame: 1 year
Reporting Status: Not Posted

4. Secondary Outcome: COPD Exacerbations Requiring Antibiotics or Corticosteroids
Time Frame: 1 year
Reporting Status: Not Posted

5. Secondary Outcome: All Cause Mortality
Time Frame: 1 year
Reporting Status: Not Posted

6. Primary Outcome: Hospitalization or ED Visit for COPD (Mean Cumulative Frequency)
Time Frame: 1 yr
Measure: Mean (95% Confidence Interval); unit: events per year
Arm/Group | Disease Management for COPD | Usual Care
Number analyzed (Participants) | 372 | 371
events per year | 0.48 [.35 to .61] | 0.82 [.67 to .97]
Statistical Analysis 1: Comparison: Disease Management for COPD vs Usual Care; primary outcome is mean cumulative frequency of COPD related hospitlaizations and ED visits ;ver 1 yr: 0.48 for disease management; 0.82 for usual care, difference 0.34 (95% CI 0.15 to 0.52; P<0.001); Test type: Superiority or Other; p < 0.001, mean cumulative frequency

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes